CLINICAL TRIAL: NCT03001765
Title: Impact of an Intensive Monitoring Strategy in Symptomatic Patients With Suspected Arrhythmia
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Elizabeth Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPACT
Record Dates: First submitted 2016-12-16; First posted 2016-12-23 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Suspected Arrhythmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensive Monitoring Strategy: Reveal LINQ™ Insertable Cardiac (Other): Intensive monitoring strategy of discharging from the Emergency Department with an external 30 day cardiac monitoring system. A negative 30 day external monitor report will be followed by an implantable cardiac monitor.
  Interventions: Other: Intensive Monitoring Strategy: Reveal LINQ™ Insertable Cardiac Monitoring System".

INTERVENTIONS:
Other: Intensive Monitoring Strategy: Reveal LINQ™ Insertable Cardiac Monitoring System". — Intensive monitoring strategy of discharge from Emergency Department with 30 day SEEQ external monitor, followed by implantable cardiac Reveal LINQ monitor if negative 30 day result.

SUMMARY:
Hypothesis:

Patients that were previously discharged from the emergency department with a subsequent non-diagnostic 30 day external patch monitor for suspected arrhythmia will benefit from early Reveal LINQ™ Insertable Cardiac Monitoring System placement.

Primary Study Objectives:

To evaluate the outcome of an intensive monitoring strategy (patients with a negative 30 day SEEQ™ Mobile Cardiac Telemetry (MCT) System result are purposed over for a Reveal LINQ™ Insertable Cardiac Monitoring System) in patients with suspected but no previously documented arrhythmias that result in a clinically actionable event.

DETAILED DESCRIPTION:
Eligible patients will be enrolled after presentation to the Emergency Department of St. Elizabeth Healthcare with symptoms suggestive of cardiac arrhythmia and prior to leaving the emergency department. Patients will be exited from the study and considered complete at the identification of a cardiac arrhythmia as defined in the protocol (endpoint), or 12 months from enrollment date, whichever occurs first.

Protocol defined endpoints

1. Planned insertion of a permanent pacemaker, implantable cardiac defibrillator or chronic resynchronization device.
2. Planned cardiac ablation procedure.
3. Initiation of medical therapy for the purpose of treating dysrhythmia.
4. Diagnosis of arrhythmia not requiring medical or invasive arrhythmia management.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Patient present to the ED with symptoms suggestive of cardiac arrhythmia
* English is the patient's primary language
* Willing and able to provide consent for participation in the study
* Patient is willing and able to comply with the protocol including the required follow-up

Exclusion Criteria:

* Refusal to participate
* Age < 18 years of age
* Unable to provide consent
* Current implanted loop recorder, or loop recorder explanted within the past 12 months.
* Current implant of cardiac implantable electronic device, such as permanent pacemaker (PPM), implantable cardioverter defibrillator (ICD), or cardiac resynchronization therapy (CRT) device.
* Life expectancy < 12 months
* History of prior cardiac ablation or electrophysiology study for suspected arrhythmia
* Investigator decision related to serious comorbidities or identification of reversible cause
* Unable to comply with follow-up procedures
* Previous documented diagnosis of cardiac arrhythmia by holter monitor, event monitor, ECG.
* Currently taking antiarrhythmic medication for a previously documented cardiac arrhythmia
* History of or suspected diagnosis of Postural Orthostatic Tachycardia Syndrome (POTS)
* Patient has unusual thoracic anatomy that precludes proper SEEQ patch placement
* Patient is enrolled in another study that could confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects in which a cardiac arrhythmia is detected from the study intervention of an intensive monitoring strategy. | 12 months or less
  The number of subjects in which any cardiac arrhythmia that results in a clinically actionable event will be recorded. Descriptive statistics will be used to describe baseline study subject characteristics and the clinically actionable findings.
The total number of all significant arrhythmias detected in the study population. | 12 months or less
  To determine the total number of all significant arrhythmias detected in the study population with the SEEQ™ Mobile Cardiac Telemetry (MCT) System and/or the implantable Reveal LINQ™ Insertable Cardiac Monitoring System. Subjects completing each phase of the intervention will be expressed as a percentage, as well as the percent of subjects with negative findings at the end of study participation.
The average time, in days, to diagnosis of significant arrhythmia using the intervention of intensive monitoring. | 12 months or less
  Compute the average time, in days, to diagnosis of significant arrhythmia using the intensive strategy of monitoring subjects with the SEEQ™ Mobile Cardiac Telemetry (MCT) System and the Reveal LINQ™ Insertable cardiac monitor.
Identify and categorize arrhythmia subtypes using the intensive monitoring strategy. | 12 months or less
  Of those subjects with clinical findings, identify the action required, and categorize outcome as desirable, undesirable, or inconclusive.

SECONDARY OUTCOMES:
Evaluate if the intensive monitoring strategy causes a reduction in the number and overall expense of ancillary diagnostic testing used to aid in the detection of suspected cardiac arrhythmias. | 12 months or less
  In subjects with recurrent symptom, compare the intensive strategy to the number of prior tests that have been performed. In subject who have previously presented with symptoms and undergone prior diagnostic evaluation, estimate the total expense of all prior evaluation and diagnostic testing performed.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Carrigan, MD, FHRS, Principal Investigator — St Elizabeth Healthcare
Locations (1):
- St. Elizabeth Healthcare, Edgewood, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.